CLINICAL TRIAL: NCT06680908
Title: Investigating the Effects of Combined Mental and Physical Stress
Brief Title: Impact of Combined Stress on Biomarkers of Stress
Status: Completed | Type: Observational
Sponsor: Texas State University (Other)
Collaborators: Texas State University, San Marcos (Other)
Responsible Party: Principal Investigator, Matt McAllister, Associate Professor, Texas State University
Other Study IDs: Combined Stress
Record Dates: First submitted 2024-11-06; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Physiological Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — the participants collected their own saliva using the passive drool method. Each sample was collected by allowing saliva to pool in mouth, by tilting their head forward and gently guiding saliva into a tube. Each sample was approximately .1 tbsp (1.5mL) of saliva.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dual stress challenge group: VR-ASD & Exercise test: VR-ASD:
  ~90 second VR scenario, subject was instructed that they are a responding officer to an active shooter, and they must find and eliminate the shooter. They then must walk down a 10 foot hallway, find the shooter, and take them out with their Glock 17 training pistol.
  Exercise Test:
  30 squats in 45 seconds, tempo set by metronome at 80bpm. Each rep must consist of 90 degree knee flexion with their back straight. Following, the subject then does 2 sets of 20 jump ropes.
- Exercise Test only: Exercise Test:
  30 squats in 45 seconds, tempo set by metronome at 80bpm. Each rep must consist of 90 degree knee flexion with their back straight. Following, the subject then does 2 sets of 20 jump ropes.

SUMMARY:
The goal of this clinical trial is to examine the effects of combined mental and physical stress on biomarkers of stress in healthy college aged individuals. The mental stress performed is a virtual reality active shooter drill that lasts ~3 minutes, and the physical stressor is a Ruffier squat test accompanied with jump rope, in order to examine the effects of combined stress versus physical stress alone. The main question to answer is:

- What is the impact of combined stress in comparison to a single stressor on markers of subjective and biological stress?

DETAILED DESCRIPTION:
This study randomly assigned subjects to 2 groups; group one was assigned to experience the Ruffier squat test and jump rope, a physical stressor, alone. While group two was assigned to a dual stressor, the Ruffier squat test and jump rope, followed by the virtual reality active shooter drill (VR-ASD). The stress tasks marked the midway point in the study, prior to and following the stress task, researchers collected heart rate (HR), state inventory assessment (SAI), and a salivary sample in order to assess differences in perceived and physiological stress levels.

All procedures from this project were reviewed and approved by the University Institutional Review Board.

The experimental procedures began upon arrival to the testing site where the subjects read and signed the informed consent document, had their body composition measurements taken by the inbody, as well as height taken, they were then exported to the gymnasium where they were instructed to rinse their mouth with water and rest. There was 4 collection periods in this study, where a SAI, HR, and saliva sample was taken; 1) 30 minutes pre exercise test 2) immediately pre exercise test 3) 5 minutes post exercise test 4) 30 minutes post exercise.

Virtual Reality- Active Shooter Drill (VR-ASD):

The VR-ASD is a virtual reality simulation that required the subject to wear a VR headset, carry a Glock 17 training pistol, and navigate the VR environment by physically moving on their own without interruption. The VR was performed in an open gymnasium, much larger than the scenario, to allow for ample room to roam the scenario. Following a familiarization period, the subject is then told they are a responding officer to an active shooter where they will be asked to find and eliminate the target. The subject then physically walked down a 10-foot hallway in VR where they encountered 2 victims of the shooting. One of the victims has traumatic injuries, while the other victim runs out of the room with the shooter with gunshot wounds to their arm and leg. Once the subject reaches the room with the shooter, they will observe a victim with a traumatic head injury, and the shooter firing his handgun at the last victim. If the subject hadn't fired their weapon at this point, the shooter would then begin open firing at the participant. Once the shooter had been shot by the participant, the shooter fell to the ground and the scenario ended.

Exercise test:

The participants performed 30 squats in 45 seconds with a tempo set by a metronome at 80 bpm. Each repetition consisted of squatting down to 90-degree knee flexion and back up with their back straight and arms extended in front. Failure to meet 90 degree flexion after two warnings resulted in disqualification and they were not be able to continue the exercise intervention due to not meeting the criteria. The squat test is completed in 3 minutes. The participants sat for five minutes before having their resting HR recorded, they then performed the 30 squats and had their HR recorded immediately following, then waited 60 seconds before getting their final HR recording to complete the squat test. Following, they were then instructed to perform 2 sets of 20 jump ropes under 90 seconds.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy, aged 18-39
* free from any known cardiovascular or metabolic diseases,
* free from any major stressors within the last 30 days such as birth of a child, abortion, or divorce.

Exclusion Criteria:

* subjects are required to not have a history of motion sickness, or vertigo
* not previously diagnosed with a brain injury or epilepsy, asthma, or currently taking psychological medication

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects who participated were 18-39, healthy, college aged students recruited from Texas State University campus.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-05-04 (Actual); Study Completion 2024-05-04 (Actual)

PRIMARY OUTCOMES:
Salivary secretory IgA | Up to 6 months
  SIgA is a marker of immune function and salivary SIgA concentrations tend to increase when exposed to stress
Salivary alpha amylase | Up to 6 months
  salivary alpha amylase is an enzyme involved in digestive processes. Amylase concentration in saliva have been shown to reflect sympathetic stress. Thus, as sympathetic stress increases, salivary amylase concentrations tend to increase.
Heart Rate | Up to 6 months
  heart rate reflects activity from parasympathetic and sympathetic nervous system and increases when exposed to stress
State Anxiety Inventory | Up to 6 months
  state anxiety inventory is a subjective scale which includes six short statements such as "I feel calm" or "I feel tense" and composite scores of participant responses are used for analysis. Higher values reflect higher subjected anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas State Univeristy, San Marcos, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Consent was not obtained for data sharing.